CLINICAL TRIAL: NCT00823771
Title: A Pilot Study in the Transfer of Follow-up Reviews to the General Practitioner for Prostate Cancer Patients Who Have Undergone Radiotherapy Treatment
Brief Title: A Pilot Study to Assess the Follow-up of Prostate Cancer Patients Who Have Undergone Radiotherapy Treatment
Acronym: PROFUGO
Status: Terminated | Type: Observational
Why Stopped: Data review showed that the study was underpowered to draw clear conlcusions
Sponsor: Barwon Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: ALCC 07.01
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2013-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Reviewed by radiation oncologist
- Reviewed by general practitioner

SUMMARY:
This is a pilot study assessing the role of the general practitioner in performing follow-up reviews on men who have recently completed radical radiotherapy for prostate cancer. This will be measured primarily by assessing any changes to the patient's health-related quality of life which will be evaluated by the completion of questionnaires by the participant at each review visit. The study aims to confirm that patient outcome is identical, independent of whether follow-up is performed by a specialist or the patient's General Practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Men with a tumour T1-3 stage prostate cancer and have had radical radiotherapy with curative intent
* Are between six and twelve months post-treatment completion
* Have completed all treatment for prostate cancer (including hormonal deprivation therapy)
* Have no evidence of metastatic disease
* ECOG performance status of between 0-1
* Remains willing to comply with study requirements
* Has maintained contact with an individual general practitioner

Exclusion Criteria:

* Persistent complications resulting from treatment defined as a minimum Grade 3 treatment toxicity
* Unable to complete self-administered questionnaires
* Are currently enrolled in a study that requires specialist follow-up
* Life expectancy of less than 6 months
* Surgery to remove the prostate
* Evidence of biochemical failure

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men approximately six months post-completion of radical radiotherapy treatment for prostate cancer who have not experienced significant treatment toxicities or disease progression.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2007-10; Primary Completion 2012-10 (Actual); Study Completion 2014-04-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the patient's health-related quality of life that will be assessed by the patient completing self-administered questionnaires | QOL questionnaires will be asked to be completed at baseline, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54 and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Lynch, BMedSc, MBBS, Principal Investigator — Barwon Health
Locations (1):
- Andrew Love Cancer Centre, Geelong, Victoria, Australia